CLINICAL TRIAL: NCT00073957
Title: Zevalin And Rituxan For The Treatment Of Relapsed Or Refractory Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Brief Title: Y 90 Ibritumomab Tiuxetan &Rituximab Relapsed or Refractory Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Robin Joyce, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003P000182; CDR0000341437 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Lymphoma
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Large-Cell, Anaplastic | interventions — Rituximab; Cytarabine; ibritumomab tiuxetan

STUDY DESIGN:
Intervention Model Description: Standard Phase 2
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Y-90 Ibritumomab Tiuxetan (Experimental): Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab and central nervous system prophylaxis with Cytarabine or liposomal cytarabine
  Interventions: Biological: rituximab; Drug: cytarabine; Drug: liposomal cytarabine; Radiation: yttrium Y 90 ibritumomab tiuxetan

INTERVENTIONS:
Biological: rituximab
  Other Names: Rituxan
Drug: cytarabine — to be used for CNS prophylaxis
  Other Names: cytosine arabinoside
Drug: liposomal cytarabine — to be used as CNS prophylaxis
  Other Names: Depocyte
Radiation: yttrium Y 90 ibritumomab tiuxetan
  Other Names: Zevalin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as yttrium Y 90 ibritumomab tiuxetan and rituximab, can locate cancer cells and either kill them or deliver radioactive cancer-killing substances to them without harming normal cells. Combining yttrium Y 90 ibritumomab tiuxetan with rituximab may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining yttrium Y 90 Ibritumomab tiuxetan with rituximab in treating patients who have relapsed or refractory diffuse large B-cell non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the best overall response in patients with relapsed or refractory diffuse large B-cell non-Hodgkin's lymphoma treated with yttrium Y 90 ibritumomab tiuxetan and rituximab.
* Determine the event-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

* Radioimmunotherapy: Patients receive indium In 111 ibritumomab tiuxetan IV over 10 minutes on day 1 (for imaging only); yttrium Y 90 ibritumomab tiuxetan IV over 10 minutes on day 8; and rituximab IV over 3-4 hours on days 1, 8, 15, 22, 29, and 36.
* CNS ( central nervous system)prophylaxis: Patients receive CNS prophylaxis comprising intrathecal (IT) methotrexate or IT cytarabine on days 15, 22, 29, and 36 OR IT cytarabine (liposomal) on days 15 and 29.
* Maintenance rituximab: Patients are assessed for response at week 14. Beginning at month 6, patients with stable or responding disease receive maintenance therapy comprising rituximab IV over 3-4 hours once weekly for 4 weeks. Maintenance therapy repeats every 6 months for 2 years (total of 4 courses) in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diffuse large B-cell non-Hodgkin's lymphoma, including any of the following:

  * B-cell diffuse large cell variant
  * Immunoblastic
  * Mediastinal (thymic) large cell
  * T-cell/histiocyte-rich
  * Anaplastic large B-cell
  * Intravascular large B-cell
  * Lymphomatoid granulomatosis
* Relapsed or refractory disease after at least 1 prior chemotherapy regimen and requires further treatment

  * Relapsed disease, defined as the following:

    * Appearance of any new lesion OR increase of at least 50% in the size of a previously involved site
    * 50% increase in greatest diameter of any previously identified node greater than 1 cm in the short axis OR in the sum of the perpendicular diameter (SPD) of more than 1 node
  * Progressive disease, defined as the following:

    * 50% increase from nadir in the SPD of any previously identified abnormal node
    * Appearance of any new lesion during or at the end of therapy
* CD20-positive disease by immunohistochemistry
* Bidimensionally measurable disease

  * At least 1 lesion at least 2.0 cm by CT scan
* Less than 25% bone marrow involvement by lymphoma
* No transformed lymphoma from indolent to aggressive
* No HIV- or AIDS-related lymphoma
* No hypocellular bone marrow
* No marked reduction in bone marrow precursors of 1 or more cell lines (e.g., granulocytic, megakaryocytic, or erythroid)
* No CNS lymphoma
* Ineligible for myeloablative therapy OR refused transplantation
* Ineligible for any other open yttrium Y 90 ibritumomab tiuxetan investigational protocols

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* WHO 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Lymphocyte count no greater than 5,000/mm^3 (for patients with small lymphocytic lymphoma)
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 2.0 mg/dL

Renal

* Creatinine no greater than 2.0 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 year after study participation
* No concurrent serious nonmalignant disease or infection that would preclude study participation
* No human antimurine antibody reactivity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* No prior autologous bone marrow transplantation
* No prior peripheral blood stem cell rescue
* No prior failed stem cell collection
* Prior rituximab within the past 90 days allowed provided patient has fludeoxyglucose-avid disease that is also indium In 111 ibritumomab tiuxetan-avid disease in at least 1 lesion
* More than 2 weeks since prior filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* No prior radioimmunotherapy
* No prior external beam radiotherapy (involved field or regional) to more than 25% of active bone marrow

Surgery

* More than 4 weeks since prior major surgery (except diagnostic surgery)

Other

* Recovered from all prior therapy
* More than 4 weeks since prior therapy for lymphoma
* More than 8 weeks since prior phase II investigational drugs
* No other concurrent antineoplastic therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-12 (Actual); Primary Completion 2012-01-01 (Actual); Study Completion 2012-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Joyce, MD, Study Chair — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab: Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
Period: Overall Study
Arm/Group | Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
Number analyzed (Participants) | 25
Age, Continuous [Mean (Full Range); unit: years] | 70 [60 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Response Rate = Complete and Partial Response at 12 Weeks.
Description: Definition Nodal Masses Spleen, Liver Bone Marrow CR Disappearance of all evidence of disease Partial response Regression and no new sites ≥ 50% decrease in sum of the perpendicular dimension of up to 6 largest dominant masses; no increase in size of other nodes Stable disease Failure to attain CR/PR or Progressive disease or Relapsed disease : the appearance of any new lesion or the (a) FDG-avid or PET positive prior to therapy; PET positive at prior sites of disease and no new sites on CT or PET Any new lesion or increase by ≥ 50% of previously involved sites from nadir Appearance of a new lesion(s) > 1.5 cm in any axis, ≥ 50% increase in SPD of more than one node, or ≥ 50% increase in longest diameter of a previously identified node > 1 cm in short axis > 50% increase from nadir in the SPD of any previous lesions New or recurrent involvement Lesions PET positive if FDG-avid lymphoma or PET positive prior to therapy
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
Number analyzed (Participants) | 25
participants
  CR | 5
  PR | 3
  SD | 2
  PD | 15

2. Primary Outcome: Best Response
Description: This data is the best overall response achieved by patients by the 12 month period.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab: Y 90 Ibritumomab Tiuxetan and Rituximab
Arm/Group | Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
Number analyzed (Participants) | 25
Participants
  CR | 8
  PR | 1
  SD | 1
  PD | 15

3. Secondary Outcome: Event Free Survival
Description: the median time point at which a participants experienced and event or toxicity or progression
Time Frame: 12 months
Measure: Median (Full Range); unit: months
Groups:
- Yttrium Y 90 Ibritumomab: Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
Arm/Group | Yttrium Y 90 Ibritumomab
Number analyzed (Participants) | 25
months | 2.5 [1 to 12]

ADVERSE EVENTS:
Arm/Group | Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 17/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yttrium Y 90 Ibritumomab Tiuxetan and Rituximab (N=25)
Thrombocytopenia (Investigations) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No